CLINICAL TRIAL: NCT06696651
Title: Electrical Muscle Stimulation Effect Compared With Myofascial Release on Quality of Life in Female Fibromyalgia
Brief Title: Electrical Muscle Stimulation Effect Versus Myofascial Release on Quality of Life in Female Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Mostafa Osman, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maha-004622
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Electric Stimulation; Myofascial Release; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Diet, Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electrical Myostimulation (Experimental): twenty females will receive EMS session per week ( 20mins / week ) and following healthy diet for 6 weeks .
  Interventions: Device: Electrical myostimulation; Other: healthy diet
- Myofascial Release (Active Comparator): twenty female will receive myofascial release sessions ( 2 sessions / week) and following healthy diet for 6 weeks .
  Interventions: Device: Electronic cupping; Other: healthy diet
- Healthy diet (Active Comparator): twenty females following healthy diet only for 6 weeks.
  Interventions: Other: healthy diet

INTERVENTIONS:
Device: Electrical myostimulation — Electrical myostimulation in form of suit as in fig. Blue lines demonstrate areas of electrodes inside suit. twenty females will receive EMS session per week ( 20mins / week ) and following healthy diet for 6 weeks . 20 min = 1 min warm up, 6min upper body training, 6min lower body training, 6min core training, 1 min cooling down.
  Arms: Electrical Myostimulation
Device: Electronic cupping — Twenty females will undergo two weekly myofascial release sessions and a healthy diet for six weeks, using electronic cupping to ensure equal pressure on tender points.
  Arms: Myofascial Release
Other: healthy diet — The MedDiet diet focuses on high fat intake, primarily from extra-virgin olive oil, in vegetable dishes, and a high consumption of low-glycemic index carbohydrates like wholegrain cereals, legumes, nuts, fruits, and vegetables. Moderate to high fish consumption is also encouraged, with moderate to small amounts of poultry and dairy products. Red meat and meat products are limited or avoided.

SUMMARY:
the study was done to investigate the effect of Electrical Muscle Stimulation as muscle strengthening versus the effect of myofascial releasing on quality of life in female fibromyalgia patients while following Mediterranean diet.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain condition characterized by unrefreshing sleep, physical exhaustion, and cognitive difficulties. It affects all populations worldwide and requires a diagnosis of widespread pain for at least three months. People with Fibromyalgia show abnormal endogenous pain modulation, including reduced conditioned pain modulation and exercise-induced hypoalgesia. Exercise is considered a first-line treatment for Fibromyalgia. Electrical myostimulation has been shown to improve pain, sleep subscales, and quality of life. A potential causal link between Fibromyalgia and micronutrient deficiency has been suggested. The study focuses on fibromyalgia, which affects mostly females and is difficult to diagnose easily. Electrical myostimulation and myofascial release are effective treatments for Fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty females have diagnosed suffering from fibromyalgia syndrome.
2. Their ages will be ranged from 45 to 55 years old.
3. Their body mass index will be ranged from 25 to 34 ( overweight and obese type 1)
4. They have willingness to participate in this study.

Exclusion Criteria:

1. Peripheral vascular diseases.
2. Drug abuse.
3. Smokers.
4. Chest disease. ( either obstructive or restrictive ).
5. Clinical signs of sever cardiac events ( eg. Congestive heart disease).

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 1. Sixty females have diagnosed suffering from fibromyalgia syndrome.
  2. Their ages will be ranged from 45 to 55 years old.
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of body mass index | at baseline and after 6 weeks
  to measure body weight and height to calculate BMI for characterizing the sample.
Assessment of change of pressure pain threshold using algometry | at baseline and after 6 weeks
  Algometry is a useful tool for assessing central allodynia and hyperalgesia in FM and other pain conditions. It can provide insights into psychological factors influencing pain experience, new dynamic pain indicators, and neuroimaging techniques.

SECONDARY OUTCOMES:
assessment of fibromyalgia using Fibromyalgia Impact Questionnaire | at baseline and after 6 weeks
  The FIQ-A measures physical function, work, and well-being, including pain, fatigue, stiffness, anxiety, and depression. The Arabic version has acceptable reliability and validity criteria, suitable for clinical practice and research in the Arabic speaking population.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, new Cairo hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No